CLINICAL TRIAL: NCT03722550
Title: Growth, Safety and Efficacy of a Starter Infant Formula, Follow-up Formula, and Growing-up Milk Supplemented With a Blend of Five Human Milk Oligosaccharides: a Double-blind, Randomized, Controlled Trial
Brief Title: Second Generation Human Milk Oligosaccharides Blend Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 1624INF
Record Dates: First submitted 2018-09-27; First posted 2018-10-29 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Healthy Infants
MeSH Terms: interventions — Lactation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unique coding of the study products
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Active Comparator): Standard Starter Infant Formula, Standard Follow-up Formula, and Standard Growing-up Milk
  Interventions: Other: Standard Starter Infant Formula, Follow-up Formula, and Growing-up Milk
- Test Group 1 (Experimental): Starter Infant Formula (same as Control Group) supplemented with 1.5g/L of Human Milk Oligosaccharides, Follow-up Formula (same as Control Group) supplemented with 0.5g/L of Human Milk Oligosaccharides, and Growing-up Milk (same as Control Group) supplemented with 0.4g/L of Human Milk Oligosaccharides
  Interventions: Other: Starter Infant Formula, Follow-up Formula, and Growing-up Milk Supplemented With a Blend of Five Human Milk Oligosaccharides
- Test Group 2 (Experimental): Starter Infant Formula (same as Control Group) supplemented with 2.5g/L of Human Milk Oligosaccharides, Follow-up Formula (same as Control Group) supplemented with 0.5g/L of Human Milk Oligosaccharides, and Growing-up Milk (same as Control Group) supplemented with 0.4g/L of Human Milk Oligosaccharides
  Interventions: Other: Starter Infant Formula, Follow-up Formula, and Growing-up Milk Supplemented With a Blend of Five Human Milk Oligosaccharides
- Breastfed Group (Active Comparator): Non-randomized Breastfed reference group
  Interventions: Other: Breast-feeding

INTERVENTIONS:
Other: Starter Infant Formula, Follow-up Formula, and Growing-up Milk Supplemented With a Blend of Five Human Milk Oligosaccharides — Study formulas are administered orally, ad libitum, from enrollment until 15 months of age
  Arms: Test Group 1; Test Group 2
Other: Breast-feeding — Exclusive Breast-feeding up to 4 months of age
  Arms: Breastfed Group
Other: Standard Starter Infant Formula, Follow-up Formula, and Growing-up Milk — Standard Study formulas are administered orally, ad libitum, from enrollment until 15 months of age
  Arms: Control Group

SUMMARY:
The aim of this trial is to show that infants fed these new formulas, containing a blend of 5 Human Milk Oligosaccharides (HMOs), allow for growth in line with infants fed formulas without HMOs.

There will be different groups in the trial: three formula-fed groups and a breastfed group.

DETAILED DESCRIPTION:
These 5 HMOs are identical to the ones found naturally in human milk. They are natural prebiotics (or complex sugars) with potential health benefits. Prebiotics are natural compounds that help the establishment of beneficial gut bacteria (such as bifidobacteria), while preventing bad bacteria from doing harm. Supplementing diets with certain prebiotics has been shown to be well tolerated in adults and infants and to provide potential benefits.Therefore, the trial also aims to understand if consuming HMOs supplemented formulas could strengthen immunity and prevent common illnesses (for example, respiratory illnesses) in infants and toddlers. Furthermore, stool frequency and consistency will be monitored, so as to evaluate digestive tolerance to the formula.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of personally signed and dated informed consent document indicating that the infant's parent(s)/Legally Acceptable Representative has been informed of all pertinent aspects of the study.
2. Infants whose parent(s)/Legally Acceptable Representative have reached the legal age of majority in the countries where the study is conducted.
3. Infants whose parent(s)/Legally Acceptable Representative are willing and able to comply with scheduled visits, and the requirements of the study protocol.
4. Infants whose parent(s)/Legally Acceptable Representative are able to be contacted directly by telephone throughout the study.
5. Infants whose parent(s)/Legally Acceptable Representative have a working freezer.
6. Infants must meet all of the following inclusion criteria to be eligible for enrollment into the study:

   1. Healthy term (37-42 weeks of gestation) infant at birth.
   2. At enrollment visit, post-natal age ≥ 7 days and ≤ 21 days (date of birth = day 0, 0.25 - 0.75 months old).
   3. At enrollment, birth weight ≥ 2500g and ≤ 4500g.
   4. For formula-fed group, infants must be exclusively consuming and tolerating a cow's milk infant formula at time of enrollment and their parent(s)/Legally Acceptable Representative must have independently elected, before enrollment, not to breastfeed.
   5. For breastfed group, infants must have been exclusively consuming breast milk since birth, and their parent(s)/Legally Acceptable Representative must have made the decision to continue exclusively breastfeeding until at least 4 month of age.

Exclusion Criteria:

1. Infants with conditions requiring infant feedings other than those specified in the protocol.
2. Infants receiving complementary foods or liquids defined as 4 or more teaspoons per day or approximately 20 g per day of complementary foods or liquids at or prior to enrollment.
3. Infants who have a medical condition or history that could increase the risk associated with study participation or interfere with the interpretation of study results, including:

   1. Evidence of major congenital malformations (e.g., cleft palate, extremity malformation).
   2. Suspected or documented systemic or congenital infections (e.g., human immunodeficiency virus, cytomegalovirus, syphilis).
   3. History of admission to the Neonatal Intensive Care Unit (NICU), with the exception of admission for jaundice phototherapy.
   4. Other severe medical or laboratory abnormality (acute or chronic) which, in the judgment of the investigator, would make the infant inappropriate for entry into the study.
4. Infants who are presently receiving or have received prior to enrollment any of the following: medication(s) or supplement(s) which are known or suspected to affect the following: fat digestion, absorption, and/or metabolism (e.g., pancreatic enzymes); stool characteristics (e.g., glycerin suppositories, bismuth-containing medications, docusate, Maltsupex, or lactulose); growth (e.g. insulin or growth hormone); gastric acid secretion; or any study outcomes.
5. Currently participating or having participated in another clinical trial since birth

Ages: 7 Days to 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 789 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
To compare the growth of infants between the groups | From Study Day 1 to 4 months of age
  To compare the growth (weight gain, g/day) of infants randomized to Test Groups (TG1 or TG2) versus Control Group (CG)
To compare recurrent incidences of illness of infants between the groups | From Study Day 1 to 15 months of age
  To compare recurrent incidences of illness (specifically lower and upper respiratory tract illnesses including bronchitis/bronchiolitis), of infants randomized to Test Groups (TG1 or TG2) versus Control Group (CG)

SECONDARY OUTCOMES:
Infant illness and infection outcomes | at different stages of feeding 1st age Infant Formula, 2nd age Follow-up Formula, and 3rd age Growing-up Milk when applicable
  Specific parent-reported infant illness symptoms and physician confirmed diagnoses of lower respiratory tract infection (LRTI), upper respiratory tract infection (URTI), total respiratory tract infection (TRTI), gastrointestinal infection (GII), ear illness [including: otitis media (OM), ear infection, ear inflammation, and ear pain], and fever will be combined to report infant illness and infection outcomes (Episode, incidence, duration, severity, and recurrence)
Medication use (specifically antimicrobials and antipyretics) | From enrollment until 15 months of age
  Medication type and duration of intake will be combined to report the medication use
Absenteeism: Time away from daycare (infant) or work (parent) | From enrollment until 15 months of age
  Time away from daycare (infant) or work (parent)
Fecal microbiome composition, diversity, community type | Stool sample collected at infant age less than 0.75, 3, 6, 12, and 15 months of age (a subset of 105 infants per formula group; 90 breastfed infants)
  Fecal microbiota composition, diversity, and microbiota community type will be assessed using cutting-edge next generation sequencing technology and combined to report the Fecal microbiome
Fecal metabolic profile | Stool sample collected at infant age less than 0.75, 3, 6, 12, and 15 months of age (a subset of 105 infants per formula group; 90 breastfed infants)
  Measures of fecal metabolism will be combined to report fecal metabolic profile (fecal pH, fecal organic acids, as well as additional targeted/untargeted metabolomics and cell-based functional assays)
Markers of immune and gut health | Stool sample collected at infant age less than 0.75, 3, 6, 12, and 15 months of age (a subset of 105 infants per formula group; 90 breastfed infants)
  Fecal markers of immune and gut health will include secretory immunoglobulin A IgA [total], alpha-1 antitrypsin, and calprotectin.
Blood Markers of immune health | At 6 months of age
  Plasma and peripheral blood mononuclear cells, Extracellular in vivo and ex vivo circulating cytokine levels will be measured in plasma
Gastrointestinal tolerance | Stool sample collected at infant age less than 0.75, 3, 6, 12, and 15 months of age (a subset of 105 infants per formula group; 90 breastfed infants)
  Stool patterns (stool frequency and consistency), Gastrointestinal symptoms, Gastrointestinal-related behaviors, and milk intake will be combined to report the gastrointestinal tolerance
Cognitive and behavioral outcomes | At 15 months of age
  Assessment at 15 months through the use of the MacArthur-Bates Communicative Development Inventories (MCDI) and the Early Childhood Behavior Questionnaire (ECBQ), two parent-reported questionnaires that evaluate early language/vocabulary and development of communication skills, that will be combined to report the cognitive and behavioral outcomes
DNA Genotyping of fucosyltransferase 2 and 3 (secretor status) | At Study Day 60 +/- 5 days
  Association between secretor status and illnesses/infections via microbiome modulation will be evaluated.
Breastmilk collection for Human Milk Oligosaccharides profile analysis (breastfeeding mothers only) | At Study Day 90 +/- 5 days
  A small sample of milk (1ml) will be hand pumped, collected in an Eppendorf tube and stored frozen
Anthropometric measurements: Weight | From enrollment until 15 months of age
  Weight measurements in grams to report anthropometric measurements.
Anthropometric measurements: Length | From enrollment until 15 months of age
  Length measurements in centimeters to report anthropometric measurements.
Anthropometric measurements: Head circumference | From enrollment until 15 months of age
  Head circumference measurements in centimeters to report anthropometric measurements.
Anthropometric measurements: BMI | From enrollment until 15 months of age
  BMI measurements in kg/m^2 to report anthropometric measurements.
Anthropometric measurements: World Health Organization (WHO) growth standard calculated z-scores | From enrollment until 15 months of age
  WHO growth standard z-scores including weight-for-age, length-for-age, weight-for-length, head-circumference-for-age, BMI-for-age and weight velocity will be calculated and combined to report anthropometric measurements.
Vital signs: Infant respiration | From enrollment until 15 months of age
  Infant respiration in breaths per minute will also be measured to report vital signs
Vital signs: Heart rate | From enrollment until 15 months of age
  Heart rate in beasts per minute will also be measured to report vital signs
Vital signs: Body temperature | From enrollment until 15 months of age
  Body temperature in Celsius degree will also be measured to report vital signs
Standard adverse events (AEs) reporting for safety assessment | From the time the informed consent form has been signed at enrollment infant age less than 21 days or 0.75 months through the 2 weeks post-study telephone contact at infant age 464 days
  Reported adverse events (AEs) and Serious Adverse Events (SAEs) include type, incidence, severity, seriousness and relation to feeding
Bone index measurement | From enrollment until 15 months of age
  Bone index measurement will be conducted using a non-invasive and radiation-free ultra-sound sonometer measuring bone transmission time and speed of sound at the radius and tibia site, including also the measurement of the femur and radius length
Dietary pattern | From 6 months of age until 15 months of age
  Dietary pattern will be evaluated using a Food frequency questionnaire including sixteen key food groups for infants and young children

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander Krasnow, Lek. Med., Principal Investigator — Gdańskie Centrum Zdrowia Sp. Z o.o.; Wiesław Olechowski, Dr n.med., Principal Investigator — ALERGO-MED Specjalistyczna Przychodnia Lekarska Sp. Z o.o.; Sylwia Korzyńska, MD, Principal Investigator — Centrum Medyczne Pratia Ostrolęka; Anna Płoszczuk, Dr. n.med., Principal Investigator — Prywatna Praktyka Lekarska Gabinet Pediatryczno-Alergologiczny Anna Płoszczuk; Magdalena Sidorowicz, Dr., Principal Investigator — Centrum Medyczne Pratia Warszawa; Grażyna Jasieniak-Pinis, Lek. Med., Principal Investigator — ATOPIA Niepubliczny Zakład Opieki Zdrowotnej Poradnie Specjalistyczne; Bartosz Korczowski, PhD MD Dr, Principal Investigator — Korczowski Bartosz Gabinet Lekarski; Piotr Korbal, Dr., Principal Investigator — Szpital Uniwersytecki nr 2 Im. Dr Jana Biziela w Bydgoszczy Oddział Kliniczny Noworodków, Wcześniaków z Intensywną Terapią Noworodka wraz z; Marta Żołnowska, Lek. Med., Principal Investigator — Centrum Medyczne Plejady; Bogusław Cimoszko, Lek. Med., Principal Investigator — Clinical Vitae Sp z o.o. Poradnia Podstawowej Opieki Zdrowotnej; Wanda Furmaga-Jabłonska, Prof., Principal Investigator — Uniwersytecki Szpital Dziecięcy w Lublinie; Marzena Nowak, Dr., Principal Investigator — Centrum Medyczne PROMED; Georgios Marek Vasilopoulos, Dr., Principal Investigator — Centrum Innowacyjnych Terapii Sp. z o.o.; Viktor Bauer, MD, Principal Investigator — Dr. Kenessey Albert Kórház-Rendelőintézet; Robert Simkó, MD, Principal Investigator — Futurenest Kft.; István Laki, MD, Principal Investigator — Kanizsai Dorottya Kórház; Éva Kovács, MD, Principal Investigator — Házi Gyermekorvosi Rendelő / Babadoki Kft.; Éva Szabó, MD, Principal Investigator — Csolnoky Ferenc Kórház; István Tokodi, MD, Principal Investigator — Mentaház Magánorvosi Központ Kft.; Zsuzsanna Tengelyi, MD, Principal Investigator — Clinexpert Kft.; Katalin Fister, MD, Principal Investigator — Clinexpert Gyöngyös Egészségügyi Szolgáltató Kft.; Anton Bilev, MD, Principal Investigator — MC ''Sveti Ivan Rilski - Chudotvorets''; Miroslava Bosheva, MD, Principal Investigator — University Multiorofile Hospital for active treatment Sveti Georgi EAD, Pediatric clinic; Toni Grigorov, MD, Principal Investigator — Multiprofile Hospital for Active Treatment City Clinic - Sveti Georgi EOOD,Department of Paediatrics,; Rositsa Karcheva-Beloeva, MD, Principal Investigator — Medical Center-1-Sevlievo; Margarita Koleva, MD, Principal Investigator — Diagnostic-consultative center Ritam TR; Stelyana Kraeva, MD, Principal Investigator — Alitera -Med-Medical Center; Olga Nikolova, MD, Principal Investigator — Multiprofile Hospital for Active Treatment Sveti Ivan Rilski Kozloduy,Department of Pediatrics; Tatyana Stoeva, MD, Principal Investigator — Medical Centre - Izgrev; Irina Popova, MD, Principal Investigator — University Hospital 'Deva Maria', Department for Naonatology; Svilen Dosev, MD, Principal Investigator — Multiprofile Hospital for Active treatment Ruse AD, Department of Paediatrics; Stefan Banov, MD, Principal Investigator — SMA Dr Stefan Banov; Sirma Dimitrova, MD, Principal Investigator — Medical Center Excelsior; Malgorzata Arciszewska, MD, Principal Investigator — Poliklinika Ginekolo.-Poloznicza
Locations (34):
- Bulgaria (13):
  - Sveti Ivan Rilski - Chudotvorets, Blagoevgrad
  - University Hospital Deva Maria, Department for Naonatology, Burgas
  - Multiprofile Hospital for Active Treatment Sveti Ivan Rilski Kozloduy,Department of Pediatrics, Kozloduy
  - Multiprofile Hospital for Active Treatment City Clinic - Sveti Georgi EOOD,Department of Paediatrics, Montana
  - University Multiorofile Hospital for active treatment Sveti Georgi EAD, Pediatric clinic, Plovdiv
  - Multiprofile Hospital for Active treatment- Ruse AD, Department of Paediatrics, Rousse
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - 1st Pediatric Consultative Clinic, Sofia
  - Medical Center Excelsior, Sofia
  - Medical Centre - Izgrev EOOD, Sofia
  - Alitera-Med-Medical Center EOOD, Sofia
  - Diagnostic-consultative center Ritam TR'' OOD, Stara Zagora
  - SMA Dr Stefan Banov, Stara Zagora
- Hungary (8):
  - Dr. Kenessey Albert Kórház-Rendelőintézet Csecsemő és Gyermekosztály, Balassagyarmat
  - Clinexpert Kft., Budapest
  - Clinexpert Gyöngyös Egészségügyi Szolgáltató Kft., Gyöngyös
  - Futurenest Kft., Miskolc
  - Kanizsai Dorottya Kórház Csecsemő és Gyermekgyógyászati Osztály, Nagykanizsa
  - Házi Gyermekorvosi Rendelő / Babadoki Kft., Szeged
  - Mentaház Magánorvosi Központ Kft., Székesfehérvár
  - Csolnoky Ferenc Kórház, Veszprém
- Poland (13):
  - Poliklinika Ginekolo.-Poloznicza, Bialystok
  - Szpital Uniwersytecki nr 2, Bydgoszcz
  - Clinical Vitae Sp z o.o. Poradnia Podstawowej Opieki Zdrowotnej, Gdansk
  - Gdańskie Centrum Zdrowia Sp. Z o.o, Gdansk
  - Centrum Medyczne Plejady, Krakow
  - Grażyna Jasieniak-Pinis ATOPIA Niepubliczny Zakład Opieki Zdrowotnej Poradnie Specjalistyczne, Krakow
  - Centrum Medyczne PROMED, Krakow
  - Uniwersytecki Szpital Dziecięcy w Lublinie, Lublin
  - Centrum Medyczne Pratia Ostrolęka, Ostrołęka
  - Centrum Innowacyjnych Terapii Sp. z o.o., Piaseczno
  - Korczowski Bartosz Gabinet Lekarski, Rzeszów
  - ALERGO-MED Specjalistyczna Przychodnia Lekarska Sp. Z o.o, Tarnów
  - Centrum Medyczne Pratia Warszawa, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bosheva M, Tokodi I, Krasnow A, Pedersen HK, Lukjancenko O, Eklund AC, Grathwohl D, Sprenger N, Berger B, Cercamondi CI; 5 HMO Study Investigator Consortium. Infant Formula With a Specific Blend of Five Human Milk Oligosaccharides Drives the Gut Microbiota Development and Improves Gut Maturation Markers: A Randomized Controlled Trial. Front Nutr. 2022 Jul 6;9:920362. doi: 10.3389/fnut.2022.920362. eCollection 2022. PMID 35873420